CLINICAL TRIAL: NCT01524224
Title: A Phase 1 Dose-Escalation Study of LY2495655, an Anti-Myostatin Monoclonal Antibody, in Patients With Advanced Cancer
Brief Title: A Dose-Escalation Study in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 11207; I1Q-MC-JDDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-01

CONDITIONS: Advanced Cancer
Keywords: Metastases; Neoplasm; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — landogrozumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2495655 (Experimental): Administered intravenously (IV) every 2 weeks (14 days) for four (4) 14 day cycles. Participants receiving clinical benefit may continue to receive treatment until one or more of the discontinuation criteria are met.
  Starting dose in Part 1 (dose escalation) will be 2 mg. The dose will be subsequently increased to 7 mg, 21 mg, 70 mg, 210 mg, and 700 mg. The dose administered in Part 2 (dose confirmation) will be determined from Part 1.
  Interventions: Drug: LY2495655

INTERVENTIONS:
Drug: LY2495655 — administered intravenously

SUMMARY:
This study is a multicenter, open-label, dose-escalation phase 1 study of intravenous (IV) LY2495655 in participants with advanced cancer.

DETAILED DESCRIPTION:
This study will consist of the following parts:

1. Dose Escalation - Cohorts of at least 3 participants will be treated with increasing doses of LY2475655 until maximum tolerated dose (MTD) criteria are met in 1 of the 6 dose levels, or the 6th cohort is completed without meeting maximum tolerated dose criteria.
2. Dose Confirmation - Up to 10 more participants will be enrolled to the MTD dose level, or if it was not possible to define the MTD during dose escalation, all clinical and bioanalytical data will be reviewed to select the recommended Phase 2 dose and an up to 10 additional participants will be enrolled to this dose level.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with child bearing potential must have had a negative serum pregnancy test less than or equal to 7 days prior to the first dose of study drug
* Have an estimated life expectancy of greater than 12 weeks
* Have a histological or cytological diagnosis of cancer (with the exception of breast or prostate cancer) that is advanced and/or metastatic, for which no proven effective therapy exists or the participant has declined anticancer therapy OR
* Have a histological or cytological diagnosis of metastatic breast or metastatic prostate cancer and receiving stable anti-hormone therapy for at least 2 months
* Have adequate hematologic, hepatic, and renal function
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, or any other investigational therapy, for at least 30 days (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment and have recovered from the acute effects of therapy. Participants receiving anti-hormone therapy as specified in criteria above are not excluded

Exclusion Criteria:

* Have received treatment within 30 days of the initial dose of study drug with a drug that has not received regulatory approval for any indication
* Have serious preexisting medical conditions other than their cancer (at the discretion of the investigator)
* Have central nervous system malignancy or metastasis (screening not required)
* Have a history of severe chronic diseases that could interfere with either strength evaluation or body mass assessment during participation in this study including, but not limited to, ischemic disease (affecting the heart, brain, or extremities), uncontrolled hypertension, uncontrolled pain, severe chronic obstructive pulmonary disease, uncompensated heart failure (New York Heart Association Class III or IV), uncontrolled diabetes, or liver cirrhosis (Child-Pugh Class C)
* Have a history of inherited or acquired neuromuscular diseases including multiple sclerosis, muscular dystrophies, or myasthenia gravis
* Have active systemic inflammatory conditions including rheumatoid arthritis, dermatomyositis, severe arthrosis, or scleroderma
* Have unstable bone lesions, or any bone instability, fusion, arthroplasty, tendon repair, synovectomy, and so on, due to any of the before-mentioned conditions or due to accident that could interfere with completion of the physical tests in this protocol
* Have chronic glucocorticosteroid use greater than 10 mg of prednisone per day or equivalent
* Have known positive test results for hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb). Screening is not required
* Have untreated hypothyroidism or hyperthyroidism
* Have history of seizures, convulsions (except previous febrile convulsions), or stroke
* Present with evidence of major depressive disorder, or history of obsessive compulsive disorder, significant psychiatric disease such as schizophrenia, bipolar disorder, or delirium
* Have depressive symptoms associated with their cancer that require treatment with any of the excluded drugs listed in protocol
* Have a previous history of discontinuation of a monoclonal antibody therapy due to allergy or severe infusion reaction
* Are scheduled to start or already receive any anti-cancer hormone treatments for breast or prostate cancer in the adjuvant or neoadjuvant setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 2 mg LY2495655: 2 milligrams (mg) LY2495655 2 milligrams (mg) every 2 weeks. Dose Escalation Phase
- 7 mg LY2495655: 7 mg LY2495655 every 2 weeks. Dose Escalation Phase
- 21 mg LY2495655: 21 mg LY2495655 every 2 weeks. Dose Escalation Phase
- 70 mg LY2495655: 70 mg LY2495655 every 2 weeks. Dose Escalation Phase
- 100 mg LY2495655: 100 mg LY2495655 every 2 weeks. Dose Confirmation Phase
- 210 mg LY2495655: 210 mg LY2495655 every 2 weeks. Dose Escalation Phase
- 300 mg LY2495655: 300 mg LY2495655 every 2 weeks. Dose Confirmation Phase
- 700 mg LY2495655: 700 mg LY2495655 every 2 weeks. Dose Escalation Phase
Period: Overall Study
Arm/Group | 2 mg LY2495655 | 7 mg LY2495655 | 21 mg LY2495655 | 70 mg LY2495655 | 100 mg LY2495655 | 210 mg LY2495655 | 300 mg LY2495655 | 700 mg LY2495655
Started | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 6
Received at Least One Dose of Study Drug | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 6
Completed | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0
Not Completed | 3 | 1 | 2 | 2 | 4 | 2 | 3 | 6
Not completed — Progressive Disease | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 5
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants that received at least one dose of study drug.
Groups:
- 2 mg LY2495655: 2 mg LY2495655 every 2 weeks. Dose Escalation Phase
- Total: Total of all reporting groups
Arm/Group | 2 mg LY2495655 | 7 mg LY2495655 | 21 mg LY2495655 | 70 mg LY2495655 | 100 mg LY2495655 | 210 mg LY2495655 | 300 mg LY2495655 | 700 mg LY2495655 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 6 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (9.2) | 78.1 (5.9) | 75.9 (3.6) | 67.1 (7.8) | 62.9 (12.5) | 78.8 (7.2) | 70.7 (7.3) | 67.9 (9.6) | 71.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 9
  Male | 1 | 3 | 2 | 3 | 3 | 3 | 1 | 4 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 3 | 2 | 3 | 3 | 3 | 3 | 6 | 25
  African | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Hispanic | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-related Adverse Events
Description: A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section. An AE is summarized if the onset date is on or after the first dose of study drug and within 30 days after the last dose, or it occurred before the first dose of study drug and worsened while on the therapy.
Time Frame: Baseline through End of Study (up to 51 months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 mg LY2495655 | 7 mg LY2495655 | 21 mg LY2495655 | 70 mg LY2495655 | 100 mg LY2495655 | 210 mg LY2495655 | 300 mg LY2495655 | 700 mg LY2495655
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 4 | 3 | 3 | 6
Participants | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve From Time 0 to 336 Hours (AUC[0-336]) of LY2495655
Description: AUC(0-336h) is the area under the drug concentration versus time curve within a dosing interval (0-336 hours). Due to the small number per cohort (participants dropping out) calculations of the accumulation factor of exposure for repeated every-other-week dosing were based on simulated area under the drug concentration versus time curve within a dosing interval (AUCτ) instead of observed values. The 90-percentage confidence interval was calculated as the predictive interval.
Time Frame: Cycle 1 and Cycle 4 Days 1 (pre-dose, end of infusion, 2hr, 6hr, 10-12hr after the infusion ends) and Day 2, 3, 5, 8
Population: All participants who received at least one dose of study drug and had evaluable pharmacokinetic data. Confidence Interval calculated as predictive interval and summarized from simulated PK profiles in 1000 virtual participants for each dose using a population PK model for LY2495655.
Measure: Median (90% Confidence Interval); unit: micromolar*hr (µM*hr)
Arm/Group | 2 mg LY2495655 | 7 mg LY2495655 | 21 mg LY2495655 | 70 mg LY2495655 | 100 mg LY2495655 | 210 mg LY2495655 | 300 mg LY2495655 | 700 mg LY2495655
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3
micromolar*hr (µM*hr)
  Cycle 1 | 0.426 [0.309 to 0.605] | 1.62 [1.18 to 2.35] | 5.36 [3.87 to 7.94] | 19.5 [13.8 to 28.7] | 28.2 [20.2 to 41.6] | 60.4 [43.2 to 89.4] | 86.8 [62.1 to 128] | 204 [146 to 302]
  Cycle 4 | 0.622 [0.408 to 0.931] | 2.63 [1.63 to 4.05] | 10.0 [6.00 to 15.3] | 39.2 [23.1 to 61.0] | 57.6 [33.9 to 89.8] | 124 [73.4 to 195] | 179 [106 to 280] | 424 [252 to 660]

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2495655
Time Frame: Cycle 1 and Cycle 4 Days 1 (pre-dose, end of infusion, 2hr, 6hr, 10-12hr after the infusion ends) and Day 2, 3, 5, 8
Population: All participants who received at least one dose of study drug and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | 2 mg LY2495655 | 7 mg LY2495655 | 21 mg LY2495655 | 70 mg LY2495655 | 100 mg LY2495655 | 210 mg LY2495655 | 300 mg LY2495655 | 700 mg LY2495655
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3
nanomolar (nM)
  Cycle 1 | 6.58 (7) | 11.5 (12) | 38.3 (20) | 101.0 (12) | 754.0 (37) | 221.0 (8) | 1360.0 (27) | 392.0 (14)
  Cycle 4: number analyzed (Participants) | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 3
  Cycle 4 | 6.67 (NA) — CV% not calculated when n=2. Individual parameter (7.74, 5.75). | 12.6 (9) | 60.2 (NA) — CV% not calculated when n=2. Individual parameter (55.62, 65.11). | 165.0 (16) | 1020.0 (NA) — CV% not calculated when n=2. Individual parameter (768.76, 1349.52). | 307.0 (24) | 2010.0 (31) | 559.0 (18)

ADVERSE EVENTS:
Arm/Group | 2 mg LY2495655 | 7 mg LY2495655 | 21 mg LY2495655 | 70 mg LY2495655 | 100 mg LY2495655 | 210 mg LY2495655 | 300 mg LY2495655 | 700 mg LY2495655
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 1/3 | 1/4 | 2/3 | 1/3 | 2/6
Other Adverse Events (participants affected / at risk) | 2/4 | 3/3 | 3/3 | 3/3 | 4/4 | 2/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY2495655 (N=4) | 7 mg LY2495655 (N=3) | 21 mg LY2495655 (N=3) | 70 mg LY2495655 (N=3) | 100 mg LY2495655 (N=4) | 210 mg LY2495655 (N=3) | 300 mg LY2495655 (N=3) | 700 mg LY2495655 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 mg LY2495655 (N=4) | 7 mg LY2495655 (N=3) | 21 mg LY2495655 (N=3) | 70 mg LY2495655 (N=3) | 100 mg LY2495655 (N=4) | 210 mg LY2495655 (N=3) | 300 mg LY2495655 (N=3) | 700 mg LY2495655 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (18) | 0 (0) | 1 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (31) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (3) | 1 (2) | 1 (10) | 3 (6) | 0 (0) | 2 (8) | 1 (5)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (13) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (4) | 1 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (17)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (19) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (6) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (9) | 1 (23) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (16)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (19)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (17)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (18) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 1 (19)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (6) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days